CLINICAL TRIAL: NCT01599949
Title: A Phase 2, Multicenter, Single-Arm, Study to Evaluate the Efficacy and Safety of Single-Agent Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib, in Subjects With Mantle Cell Lymphoma Who Progress After Bortezomib Therapy
Brief Title: A Study to Evaluate the Efficacy and Safety of Ibrutinib, in Patients With Mantle Cell Lymphoma Who Progress After Bortezomib Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100847; PCI-32765MCL2001 (Other: Janssen Research & Development, LLC); 2012-000711-88 (EudraCT Number)
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; Ibrutinib; Bruton's tyrosine kinase inhibitor; Rituximab; Bortezomib
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibrutinib (Experimental)
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Type=exact number, unit=mg, number=560, form=capsule, route=oral use. 560 mg oral ibrutinib is to be administered once daily continuously until disease progression, unacceptable toxicity, or study end, whichever occurs first. Doses can be held or reduced based on the severity of and the recovery from side effects of the study drug.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ibrutinib in patients with mantle cell lymphoma who received at least 1 prior rituximab-containing chemotherapy regimen and who progressed after bortezomib therapy.

DETAILED DESCRIPTION:
This is a single-arm (all patients will receive the study drug) study to evaluate the efficacy and safety of ibrutinib in patients with mantle cell lymphoma (MCL) who have received at least 1 rituximab-containing chemotherapy regimen and who progressed after bortezomib therapy. Approximately 110 eligible patients will be enrolled. During the treatment phase, patients will receive 560 mg of ibrutinib by mouth once daily continuously until disease progression, unacceptable toxicity, or study end, whichever occurs first. Treatment will be continuous (without interruption) and self-administered at home. Doses can be held or reduced based on the severity of and the recovery from side effects of the study drug. The sponsor will ensure that patients benefiting from treatment with ibrutinib will be able to continue treatment after the end of the study. Data will be collected on disease response to the treatment, on progression-free survival, overall survival, and subsequent anti-MCL therapies. Serial pharmacokinetic (study of what the body does to a drug) samples will be collected as detailed in the protocol. Safety will be monitored throughout the study. An interim analysis of the pharmacokinetic data will occur approximately 3 months after the scheduled pharmacokinetic sampling in Cycles 1 and 2 has been completed. Data will be analyzed 1 year after the last patient is enrolled for the primary analysis and 2 years after last patient is enrolled for the final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of confirmed mantle cell lymphoma (MCL) with at least 1 measurable site of disease according to Revised Response Criteria for Malignant Lymphoma
* Must have received at least 1 prior rituximab-containing chemotherapy regimen, but no more than 5 prior regimens
* Must have received at least 2 cycles of bortezomib therapy (single-agent or in combination) and have documented progressive disease during or after bortezomib therapy
* Eastern Cooperative Oncology Group performance status score 0, 1, or 2
* Hematology and biochemical values within protocol-defined parameters

Exclusion Criteria:

* Prior chemotherapy within 3 weeks, nitrosoureas within 6 weeks, therapeutic anticancer antibodies within 4 weeks, radio- or toxin-immunoconjugates within 10 weeks, radiation therapy or other investigational agents within 3 weeks, or major surgery within 4 weeks of the first dose of study drug
* Prior treatment with ibrutinib or other Bruton's tyrosine kinase inhibitors
* More than 5 prior lines of therapy (separate lines of therapy are defined as single or combination therapies that are either separated by disease progression or by a >6 month treatment-free interval
* Known central nervous system lymphoma
* Diagnosed or treated for malignancy other than MCL, except malignancy treated with curative intent and with no known active disease present for >=3 years before the first dose of study drug and felt to be at low risk for recurrence by the treating physician, adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, or adequately treated cervical carcinoma in situ without evidence of disease.
* History of stroke or intracranial hemorrhage within 6 months prior to the first dose of study drug
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists
* Requires treatment with strong CYP3A4/5 inhibitors
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Known history of human immunodeficiency virus or active infection with hepatitis C virus or hepatitis B virus or any uncontrolled active systemic infection
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 1 year after the last patient is enrolled

SECONDARY OUTCOMES:
Overall survival rate | 1 year after the last patient is enrolled and 2 years after the last patient is enrolled
Progression-free survival rate | 1 year after the last patient is enrolled and 2 years after the last patient is enrolled
Mean change from baseline in the Lym subscale | 1 year after the last patient is enrolled and 2 years after the last patient is enrolled
Mean change from baseline in the EQ-5D-5L index | 1 year after the last patient is enrolled and 2 years after the last patient is enrolled
Mean plasma concentrations of ibrutinib | Up to Cycle 2, Day 21
Maximum observed plasma concentration of ibrutinib | Up to Cycle 2, Day 21
Minimum observed plasma concentration of ibrutinib | Up to Cycle 2, Day 21
Area under the plasma concentration-time curve from time 0 to 24 hours of ibrutinib | Up to Cycle 2, Day 21
The number of participants affected by an adverse event | Up to 30 days after the last dose of study medication
Overall response rate | 1 year after the last patient is enrolled and 2 years after the last patient is enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (56):
- United States (32):
  - La Jolla, California
  - Los Angeles, California
  - Stanford, California
  - Norwalk, Connecticut
  - Jacksonville, Florida
  - Chicago, Illinois
  - Peoria, Illinois
  - Goshen, Indiana
  - Iowa City, Iowa
  - Sioux City, Iowa
  - Westwood, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Jefferson City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Hackensack, New Jersey
  - New York, New York
  - Syracuse, New York
  - Watertown, South Dakota
  - Nashville, Tennessee
  - Houston, Texas
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Morgantown, West Virginia
  - Madison, Wisconsin
- Belgium (2):
  - Bruges
  - Ghent
- France (5):
  - Grenoble
  - Mulhouse
  - Nantes
  - Pessac
  - Vandœuvre-lès-Nancy
- Israel (7):
  - Afula
  - Beer Yaakov
  - Hadera
  - Haifa
  - Nahariya
  - Petah Tikva
  - Ramat Gan
- Poland (2):
  - Chorzów
  - Lodz
- San Juan, Puerto Rico
- Russia (3):
  - Nizhny Novgorod
  - Rostov-on-Don
  - Saint Petersburg
- Spain (2):
  - Barcelona
  - Salamanca
- United Kingdom (2):
  - London
  - Plymouth

REFERENCES:
- See also: A Phase 2, Multicenter, Single-Arm Study to Evaluate the Efficacy and Safety of Single- Agent Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib, in Subjects With Mantle Cell Lymphoma Who Progress After Bortezomib Therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=3515&filename=CR100847_CSR.pdf